CLINICAL TRIAL: NCT04936503
Title: Support for the Resumption of Training of High-level Athletes Post-epidemic COVID-19
Acronym: ASCCOVID19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2020/16
Record Dates: First submitted 2021-06-02; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: COVID-19; Myocarditis
Keywords: myocardial scars; MRI; Ventricular arrhythmia; Sudden cardiac death; High-level athletes
MeSH Terms: conditions — COVID-19; Myocarditis; Death, Sudden, Cardiac | interventions — Exercise Test; Surveys and Questionnaires; Blood Specimen Collection; Biological Specimen Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-level athletes (Experimental): High level athletes are rugby players, intervention unit agents of the National Police, sports students.
  Definition of a COVID-19 positive subject : Any subject whose serology is positive (IgM and/or IgG) and/or the Reverse Transcription Polymerase Chain Reaction (RT-PCR) result is positive and/or the questionnaire is positive and/or a new electrocardiogram (ECG) abnormality.
  The COVID-19 negative subjects do not meet the definition of COVID-19 positive subjects.
  Interventions: Diagnostic Test: Resting electrocardiogram; Diagnostic Test: Stress test; Diagnostic Test: Cardiac echocardiography; Diagnostic Test: Cardiac rhythm monitoring; Other: Questionnaire; Device: Injected Cardiac MRI; Biological: Blood sampling for biobank

INTERVENTIONS:
Diagnostic Test: Resting electrocardiogram — An ECG at rest is performed for all participants at Day 0. A centralized reading is performed by one of the 6 expert cardiologists participating in the research.
Diagnostic Test: Stress test — In case of positive COVID-19 serology and/or positive COVID-19 RT-PCR and/or new ECG abnormality and/or positive questionnaire, a stress test is performed.
Diagnostic Test: Cardiac echocardiography — In case of positive COVID-19 serology and/or positive COVID-19 RT-PCR and/or new ECG abnormality and/or positive questionnaire, a Cardiac echocardiography is performed.
Diagnostic Test: Cardiac rhythm monitoring — In case of positive COVID-19 serology and/or positive COVID-19 RT-PCR and/or new ECG abnormality and/or positive questionnaire, a Cardiac rhythm monitoring is performed.
Other: Questionnaire — To determine the rhythmic risk of athletes
Device: Injected Cardiac MRI — High resolution MRIs is performed on 200 athletes :
  * 100 athletes without rhythmic abnormalities (50 individuals with positive COVID-19 status and 50 individuals with negative COVID-19 status)
  * 100 athletes with rhythmic abnormalities (50 individuals with positive COVID-19 status and 50 individuals with negative COVID-19 status)
Biological: Blood sampling for biobank — For all athletes included at the D0 inclusion visit, a centralized COVID-19 serology is performed to search for biomarkers associated with the occurrence of myocardial fibrosis: analysis of genetic determinants in relation to cardiac damage.
  For athletes who have performed MRI: Search for biomarkers associated with the occurrence of myocardial fibrosis: analyses of low-grade inflammation markers (cytokine assay and fibrosis markers).

SUMMARY:
As of March 2020, COVID-19 has become a global pandemic, halting athletic competition worldwide.

Reports from China show a high prevalence of cardiac involvement in patients with severe SARS-CoV-2 infection. These cardiac forms were found to be closely associated with adverse outcomes. The use of Magnetic resonance Imaging (MRI) had allowed to show that cardiac dysfunction could be mediated by myocardial inflammation (i.e. myocarditis). The direct implication of the virus was demonstrated with Severe Acute Respiratory Syndrome (SARS)-CoV-2 being detected on myocardial biopsies in a patient with severe heart failure.

The experience with other viruses causing acute myocarditis shows that there is a high rate of undetected injuries. Indeed, although severe heart failure can be present at the acute stage, acute viral myocarditis is most commonly pauci or asymptomatic, but still leaving occult myocardial scars visible on MRI, and exposing to higher risks of ventricular arrhythmia and sudden cardiac death over the long term.

Although athletes are younger and have fewer comorbidities than the general population and therefore are at lower risk for severe disease or death, there is a critical and urgent need to assess the prevalence of occult scars in the population of high-level athletes returning to training after the SARS-CoV-2 pandemia.

ELIGIBILITY:
Inclusion Criteria:

* High level athlete,
* Of both sexes and age ≥ 18 years,
* Affiliated to or beneficiary of a social security system,
* Free, informed, written consent signed by the participant and the investigating physician (no later than the day of inclusion and before any examination required by the research),
* Effective method of contraception for women with childbearing capacity.

Exclusion Criteria:

* Minor,
* History of ventricular arrhythmia, myocarditis, identified coronary artery disease or documented myocardial fibrosis,
* Pregnant or breastfeeding women,
* Person unable to give informed consent,
* Person deprived of liberty by judicial or administrative decision,
* Adults subject to a legal protection measure (guardianship, curator, safeguard of justice).

Specific exclusion criteria for the MRI component (Contraindications):

* Subject with an implantable pacemaker or defibrillator, intraocular metallic foreign body, intracranial metallic clip, pre 6000 Starr-Edwards type cardiac valve prosthesis, or biomedical device such as insulin pump or neurostimulator,
* Hypersensitivity to gadolinium or to one of the excipients of the contrast product used,
* Claustrophobic subjects or those unable to remain in an immobile lying position for 30 minutes,
* Renal insufficiency with creatinine clearance of less than 30 ml/min,
* A patient whose shoulder width does not allow installation in the MRI machine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Presence of rhythmic risk markers bye the questionnaire | Day 0
  Questionnaire looking for heart palpitations, chest pain/pressure and shortness of breath.
Evaluation by resting ECG of rhythmic risk marker : repolarization disorders | Day 0
  Presence or absence of repolarization disorders
Evaluation by resting ECG of rhythmic risk marker : inverted T waves | Day 0
  Presence or absence of inverted T waves
Evaluation by resting ECG of rhythmic risk marker : ST segment abnormalities | Day 0
  Presence or absence of ST segment abnormalities
Evaluation by resting ECG of rhythmic risk marker : QRS fragmentation | Day 0
  Presence or absence of QRS fragmentation
Evaluation by resting ECG of rhythmic risk marker : ventricular extrasystoles (VES) | Day 0
  Presence or absence of VES. Ventricular extrasystoles especially with short coupling (<300ms), falling on the T wave, width > 160ms, complex forms (repetitive, several morphologies, instantaneous cycle >200bpm)
Evaluation by resting ECG of rhythmic risk marker : ventricular tachycardia (VT) | Day 0
  Presence or absence of VT.
Presence of rhythmic risk markers bye the stress test | Day 0
  VES, especially with short coupling (<300ms), falling on the T wave, width > 160ms, complex shapes (repetitive, several morphologies, instantaneous cycle >200bpm), ventricular tachycardias (VT). The analysis focus on the exercise period, and the recovery period. Ventricular arrhythmias will be quantified.
Presence of rhythmic risk markers bye ECG holter | Day 0
  VES, especially with short coupling (<300ms), falling on the T wave, width > 160ms, complex shapes (repetitive, multiple morphologies, instantaneous cycle >200bpm), ventricular tachycardias (VTs). Ventricular arrhythmias are quantified.
Presence of rhythmic risk markers bye ECG monitoring during games and trainings | Day 0
  In case of moderate arrhythmia on stress test and/or Holter ECG, ECG monitoring during training sessions and matches is carried out with analysis of the tracings collected, in search of more sustained arrhythmia, particularly at the ventricular level.
Presence of rhythmic risk markers by pharmacological tests and/or electrophysiological exploration | Day 0
  If the risk is perceived as very high, pharmacological tests (Isuprel®) and/or electrophysiological exploration may be performed during hospitalization, in search of dangerous rhythm disorders, particularly at the ventricular level.

SECONDARY OUTCOMES:
Presence of myocardial fibrosis by injected MRI | Month 3
  In order to compare the prevalence of myocardial fibrosis between COVID-19 positive and COVID-19 negative individuals in high level athletes with or without rhythmic risk, a high resolution MRI is performed. The examinations is performed on 1.5 or 3T MRI systems equipped with specific antennas for cardiology. The sequence used to detect occult scars is a late enhancement sequence performed at least 15 minutes after injection of gadolinium salts, using a free-breathing 3D method, for a minimum spatial resolution of 2.5x1.25x1.25mm. The images are reviewed by a core lab at the Bordeaux University Hospital. The presence or absence of myocardial fibrosis is evaluated.
Presence of transmural localization of myocardial fibrosis by injected MRI | Month 3
  In order to compare the prevalence of myocardial fibrosis between COVID-19 positive and COVID-19 negative individuals in high level athletes with or without rhythmic risk, a high resolution MRI is performed. The examinations is performed on 1.5 or 3T MRI systems equipped with specific antennas for cardiology. The sequence used to detect occult scars is a late enhancement sequence performed at least 15 minutes after injection of gadolinium salts, using a free-breathing 3D method, for a minimum spatial resolution of 2.5x1.25x1.25mm. The images are reviewed by a core lab at the Bordeaux University Hospital. The presence or absence of transmural localization is evaluated.
Measurement of cardiac scar size by injected MRI | Month 3
  In order to compare the prevalence of myocardial fibrosis between COVID-19 positive and COVID-19 negative individuals in high level athletes with or without rhythmic risk, a high resolution MRI is performed. The examinations is performed on 1.5 or 3T MRI systems equipped with specific antennas for cardiology. The sequence used to detect occult scars is a late enhancement sequence performed at least 15 minutes after injection of gadolinium salts, using a free-breathing 3D method, for a minimum spatial resolution of 2.5x1.25x1.25mm. The images are reviewed by a core lab at the Bordeaux University Hospital. The size of scars is measured in milliliters (mL).
Search for constitutional genetic biomarkers | Month 5
  identification by sequencing of genetic variants that could have an impact on the occurrence of a severe form in individuals infected with SARS-CoV-2.
Research of inflammation markers | Month 5
  Th1/Th2/activation/inflammation/apoptosis markers are measured in sera by a Luminex test allowing the detection of 10 analytes with a commercial kit according to the manufacturer's instructions

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Bénard, MD, Study Chair — University Hospital, Bordeaux; Laurent Chevalier, MD, Principal Investigator — Medical Center of the Bordeaux-Mérignac Sports Clinic
Locations (21):
- France (21):
  - Training center Soyaux Angoulême XV Rugby, Angoulême
  - Training Center Stade Aurillacois, Aurillac
  - Aviron Bayonnais Rugby Pro Training Center, Bayonne
  - Union Bordeaux-Bègles training center, Bègles
  - Biarritz Olympique Pays Basque training center, Biarritz
  - Bordeaux University Hospital - CRB medical office - Hôpital du Tondu, Bordeaux
  - Bordeaux University Hospital - Service UDH - Hôpital Pellegrin, Bordeaux
  - CABCL Rugby Training Center, Brive-la-Gaillarde
  - US Carcassonne Rugby training center, Carcassonne
  - Union Sportive Colomiers Rugby training center, Colomiers
  - FC Grenoble Rugby training center, Grenoble
  - Stade Rochelais Rugby training center, La Rochelle
  - Racing92 training center, Le Plessis-Robinson
  - AS Montauban Rugby training center, Montauban
  - US Nevers Rugby training center, Nevers
  - Stade Français training center, Paris
  - Section Paloise Rugby training center, Pau
  - USAP Training Center, Perpignan
  - Training center Valence Romans Drôme Rugby, Romans-sur-Isère
  - Castres Olympique training center, Saïx
  - Stade Toulousain Rugby training center, Toulouse

REFERENCES:
- [Derived] Chevalier L, Cochet H, Mahida S, S SB, Benard A, Cariou T, Sridi-Cheniti S, Benhenda S, Doutreleau S, Cade S, Guerard S, Guy JM, Trimoulet P, Picard S, Dusfour B, Pouzet A, Roseng S, Franchi M, Jais P, Pellegrin I; ASCCOVID Investigators. Resuming Training in High-Level Athletes After Mild COVID-19 Infection: A Multicenter Prospective Study (ASCCOVID-19). Sports Med Open. 2022 Jun 25;8(1):83. doi: 10.1186/s40798-022-00469-0. PMID 35751748